CLINICAL TRIAL: NCT06043297
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single Oral Dose, Cross Over Bioequivalence Study of Two Products of Apixaban 5mg Tablets in Normal, Healthy, Adult, Human Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Two Products of Apixaban 5mg Tablets in Healthy, Adult, Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Collaborators: Yunus sancak (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 0335-21
Record Dates: First submitted 2023-09-04; First posted 2023-09-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2023-12

CONDITIONS: Antithrombic Drug
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban 5 mg Film Tablets (Experimental)
  Interventions: Drug: Apixaban 5MG
- Eliquis 5 mg Film tablets (Active Comparator)
  Interventions: Drug: Eliquis 5 mg

INTERVENTIONS:
Drug: Apixaban 5MG — Each film-coated tablet contains 5 mg apixaban
  Arms: Apixaban 5 mg Film Tablets
Drug: Eliquis 5 mg — Each film-coated tablet contains 5 mg apixaban
  Arms: Eliquis 5 mg Film tablets

SUMMARY:
To compare the bioavailability and characterize the pharmacokinetic profile of the sponsor's test product relative to that of reference product after single oral dose administration in normal, healthy, adult, human subjects under fasting condition and to assess the bioequivalence.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker, normal, healthy, adult, human volunteers between 18 and 45 years of age (both inclusive).
* Having a Body Mass Index (BMI) between 18.5 and 30.0 (both inclusive), calculated as weight in kg / height in m2 and body weight ≥ 60 kg.
* Not having significant diseases or clinically significant abnormal findings during screening, medical history, clinical examination, laboratory evaluations, 12 lead ECG, and chest X-ray recordings (posterior-anterior view).
* aPTT and PT within normal range.
* Able to understand and comply with the study procedures, in the opinion of the investigator.
* Able to give voluntary written informed consent for participation in the trial.
* In case of female subjects:

  * Surgically sterilized at least 6 months prior to study participation.
  * If of child bearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study.

And -Serum pregnancy test must be negative.

Exclusion Criteria:

* Known hypersensitivity to Apixaban or any excipients or any related drug or any substance.
* History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
* Ingestion of medicine [prescribed & over the counter (OTC) medication including herbal remedies, anticoagulants, antiplatelet agents, selective serotonin reuptake inhibitors (SSRIs) or serotoninnorepinephrine reuptake inhibitors (SNRIs), or non-steroidal anti-inflammatory medicinal products (NSAIDs) including acetylsalicylic acid, inhibitors of both cytochrome P450 3A4 (CYP3A4) and P-glycoprotein (P-gp), such as azole-antimycotics (e.g., ketoconazole, itraconazole, voriconazole and posaconazole)and HIV protease inhibitors (e.g., ritonavir) and Inducers of CYP3A4 and P-gp (e.g., rifampicin, phenytoin, carbamazepine, phenobarbital or St. John's Wort) and any vaccine (including COVID-19 vaccine)] at any time within 14 days prior to dosing of Period-I. In any such case subject selection will be at the discretion of the Principal Investigator.
* Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAIDs induced urticaria.
* CrCl value < 50 mL/min
* Rare hereditary problems of galactose intolerance, total lactase deficiency or glucose-galactose malabsorption
* A recent history of harmful use of alcohol (less than 2 years) i.e., alcohol consumption of more than 14 standard drinks per week for men and 07 standard drinks per week for women (A standard drink is defined as 360 mL of beer or 150 mL of wine or 45 mL of 40% distilled spirits, such as rum, whisky, brandy etc.), or consumption of alcohol or alcoholic product within 48 hours prior to receiving study medicine of Period-I.
* Smokers or who have smoked within last 06 months prior to start of the study.
* The presence of clinically significant abnormal laboratory values during screening.
* Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.
* History or presence of seizure or psychiatric disorders.
* A history of difficulty with donating blood.
* Donation of blood (1 unit or 350 mL) within a period of 90 days prior to the first dose of study medication.
* Receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication**.

  ** If investigational medicinal product is received within 90 days where there is no blood loss except safety laboratory testing, subject can be included considering 10 half-lives duration of investigational medicinal product received.
* A positive hepatitis screen including hepatitis B surface antigen and/or HCV antibodies.
* A positive test result for HIV antibody (1 &/or 2).
* Consumption of grapefruit or grape fruit products within 72 hours prior to dosing of Period-I.
* Difficulty in swallowing tablets or other oral solid dosage forms.
* An unusual diet, for whatever reason (e.g., fasting, high potassium or low-sodium), for four weeks prior to receiving the study medicine in Period-I. In any such case subject selection will be at the discretion of the Principal Investigator.
* Nursing mothers (for female subjects).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Cmax | The venous blood samples will be withdrawn at pre-dose (0.000 hour) and at 0.500, 1.000, 1.500, 2.000, 2.333, 2.667, 3.000, 3.333, 3.667, 4.000, 4.333, 4.667, 5.000, 5.500, 6.000, 8.000, 10.000, 12.000, 24.000, 36.000, 48.000 and 72.000 hours
AUC0-t | The venous blood samples will be withdrawn at pre-dose (0.000 hour) and at 0.500, 1.000, 1.500, 2.000, 2.333, 2.667, 3.000, 3.333, 3.667, 4.000, 4.333, 4.667, 5.000, 5.500, 6.000, 8.000, 10.000, 12.000, 24.000, 36.000, 48.000 and 72.000 hours

SECONDARY OUTCOMES:
AUC0-∞ | The venous blood samples will be withdrawn at pre-dose (0.000 hour) and at 0.500, 1.000, 1.500, 2.000, 2.333, 2.667, 3.000, 3.333, 3.667, 4.000, 4.333, 4.667, 5.000, 5.500, 6.000, 8.000, 10.000, 12.000, 24.000, 36.000, 48.000 and 72.000 hours

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gürpınar, Study Director — Humanis Saglık
Locations (1):
- Lambda Therapeutic Research Ltd., Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: Undecided